CLINICAL TRIAL: NCT03125915
Title: Addressing Substance Use Through Couples Voluntary Counseling and Testing (CVCT)
Brief Title: Addressing Substance Use Through CVCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tyrel Starks, Associate Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R34DA036419 (NIH); R34DA036419 (NIH)
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Results first posted 2020-02-26 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Sex, Unsafe; Drug Use
Keywords: couples HIV testing; drug intervention; communication skills
MeSH Terms: conditions — Unsafe Sex | interventions — Counseling; chitinase C

STUDY DESIGN:
Intervention Model Description: The study tests two independent variables in a fully-crossed factorial design. Half of the couples complete a substance use module during their CHTC session (half do not); half view communication skills training videos (half do not).
Who Masked: Care Provider
Masking Description: Assignment to video condition is masked with respect to the care provider. The person conducting the CHTC session is unaware of whether couples have viewed the communication skills training video prior to the session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CHTC as usual (Active Comparator): Participants receive couples HIV testing and counseling following the CDC approved protocol.
  Interventions: Behavioral: Couples HIV Testing and Counseling
- CHTC + communication skills videos (Experimental): The couple views communication skills training videos together prior to participating in a CHTC session following the CDC approved protocol.
  Interventions: Behavioral: Communication skills training video; Behavioral: Couples HIV Testing and Counseling
- CHTC + substance use module (Experimental): The couple completes a CHTC session which includes the substance use calendar and structured debriefing activity. This is administered following Step 5 in the standard CDC protocol, just prior to delivery of HIV test results.
  Interventions: Behavioral: substance use module; Behavioral: Couples HIV Testing and Counseling
- CHTC + video + substance use module (Experimental): The couple views communication skills training videos together prior to participating in a CHTC session which includes administration of the substance use calendar and structured debriefing activity.
  Interventions: Behavioral: Communication skills training video; Behavioral: substance use module; Behavioral: Couples HIV Testing and Counseling

INTERVENTIONS:
Behavioral: Communication skills training video — This video includes 4 scenes of gay couples discussing issues related to HIV prevention, testing, sexual agreements, and drug use. Each scene is viewed twice. The first viewing includes common communication errors. The second viewing portrays more skillful interpersonal communication and a more adaptive resolution to the conversation.
  Arms: CHTC + communication skills videos; CHTC + video + substance use module
Behavioral: substance use module — This activity involves completion of a calendar detailing partners' substance use in the past month and a structured debriefing activity designed to facilitate the formation of couples' goals and limits around substance use.
  Other Names: drug calendar
  Arms: CHTC + substance use module; CHTC + video + substance use module
Behavioral: Couples HIV Testing and Counseling — CHTC delivered as per the CDC protocol.
  Other Names: (CHTC)

SUMMARY:
The proposed study developed and tested two adjunct components for use in Couples HIV Testing and Counseling (CHTC) with gay-male couples: a communication skills training video and a substance use agreement module. Phase I of the study involved the creation of intervention materials and Phase II was comprised of a small randomized controlled trial comparing the additive effects of the novel components to CHTC as usual.

DETAILED DESCRIPTION:
Phase I: Utilizing formative qualitative data on the correspondence of sexual agreements, drug use, and sexual risk behavior, the study team created two adjunct intervention components:

Communication skills training videos: The team produced a brief (20-minute) communication skills training video. The video includes 4 scenes in which a gay couple is depicted discussing HIV risk, sexual agreements, or drug use. The scene is viewed twice. The first viewing includes common communication errors. The second viewing portrays the use of more effective interpersonal communication and a more adaptive outcome.

Substance use agreement module: The team developed a structured activity to assist couples in clarifying their understanding and goals around substance use. The module includes the completion of a calendar detailing recent substance use and structured debriefing questions.

Phase II: A randomized controlled trial to assess the feasibility, acceptability, and preliminary efficacy of novel intervention components will be conducted. The trial involves 70 couples (n = 140 individuals). Half of the couples are randomized to complete the drug calendar (the other half do not). Half of the couples are randomized to view communication skills training videos, the other half do not. The result is four intervention conditions:

1. CHTC as usual
2. CHTC + communication skills training videos
3. CHTC + substance use module
4. CHTC + communication skills training videos + substance use calendar

Participants complete a baseline assessment (either online or in person) prior to their intervention session. All intervention sessions are completed with both members of the couple together. Follow-up assessments are completed individually online at 1, 3, and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Both members of the couple:

1. are born male and current male gender identity;
2. identify as gay, bisexual or same-sex attracted;
3. read English at 8th grade level or better;
4. have access to the Internet;
5. agree to audio and video recording of intervention sessions;

At least one member of the couple:

1. reports the use of any drug listed on the DAST-10 in the previous 30 days.
2. s identified as HIV negative during screening and baseline assessments.

   The couple
3. has been together for at least 3 months;
4. has engaged in oral or anal sex with one another in the past 3 months;

Exclusion Criteria:

1. At baseline either member of the couple reports intimate partner violence (IPV), which is defined as serious physical or sexual violence that occurs outside the context of consensual bondage or sado-masochistic sexual play, which results in concerns about safety.
2. At the first in-person meeting, staff will be empowered to deem the couple ineligible for the intervention if they identify inconsistencies between information provided in the eligibility screener and the in-person meeting (e.g., discrepancies in age or duration of relationship) or any issues that might hinder participation (e.g., attending meeting high or drunk). The couple may also be deemed ineligible if participant responses are sufficiently inconsistent to call into question the validity of their individual responses.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — participants must identify as male gender
Enrollment: 140 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyrel J Starks, PhD, Principal Investigator — Hunter College, CUNY
Locations (1):
- Hunter College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Starks TJ, Robles G, Bosco SC, Doyle KM, Dellucci TV. Relationship functioning and substance use in same-sex male couples. Drug Alcohol Depend. 2019 Aug 1;201:101-108. doi: 10.1016/j.drugalcdep.2019.04.009. Epub 2019 May 23. PMID 31203148
- [Background] Starks TJ, Doyle KM, Shalhav O, John SA, Parsons JT. An Examination of Gay Couples' Motivations to Use (or Forego) Pre-exposure Prophylaxis Expressed During Couples HIV Testing and Counseling (CHTC) Sessions. Prev Sci. 2019 Jan;20(1):157-167. doi: 10.1007/s11121-018-0892-7. PMID 29651646
- [Background] Starks TJ, Pawson M, Stephenson R, Sullivan P, Parsons JT. Dyadic Qualitative Analysis of Condom Use Scripts Among Emerging Adult Gay Male Couples. J Sex Marital Ther. 2018 Apr 3;44(3):269-280. doi: 10.1080/0092623X.2017.1359713. Epub 2017 Aug 25. PMID 28745559
- [Result] Starks TJ, Dellucci TV, Gupta S, Robles G, Stephenson R, S Sullivan P, Parsons JT. A Pilot Randomized Trial of Intervention Components Addressing Drug Use in Couples HIV Testing and Counseling (CHTC) with Male Couples. AIDS Behav. 2019 Sep;23(9):2407-2420. doi: 10.1007/s10461-019-02455-2. PMID 30887190

RESULTS

PARTICIPANT FLOW:
Period: Baseline and Intervention
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
Started | 32 | 40 | 34 | 34
Completed | 32 | 40 | 34 | 34
Not Completed | 0 | 0 | 0 | 0
Period: 1 Month Follow up
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
Started | 32 | 40 | 34 | 34
Completed | 29 | 37 | 32 | 31
Not Completed | 3 | 3 | 2 | 3
Not completed — Lost to Follow-up | 3 | 3 | 2 | 3
Period: 3 Month Follow-up
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
Started | 32 | 40 | 34 | 34
Completed | 26 | 36 | 30 | 32
Not Completed | 6 | 4 | 4 | 2
Not completed — Lost to Follow-up | 6 | 4 | 4 | 2
Period: 6 Month Follow-up
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
Started | 32 | 40 | 34 | 34
Completed | 25 | 37 | 28 | 31
Not Completed | 7 | 3 | 6 | 3
Not completed — Lost to Follow-up | 7 | 3 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module | Total
Number analyzed (Participants) | 32 | 40 | 34 | 34 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.75 (4.89) | 27.83 (7.70) | 26.50 (2.99) | 27.76 (6.07) | 27.01 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 32 | 40 | 34 | 34 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black (non-Hispanic/Latino) | 6 | 9 | 4 | 4 | 23
  Latino/Hispanic | 8 | 7 | 13 | 7 | 35
  White (non-Hispanic/Latino) | 15 | 19 | 13 | 17 | 64
  Multi-racial or Other | 3 | 5 | 4 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 32 | 40 | 34 | 34 | 140
Reported any drug use [Count of Participants; unit: Participants] | 25 | 34 | 24 | 29 | 112
Condomless sex with casual partners [Count of Participants; unit: Participants] | 9 | 8 | 8 | 4 | 29
Drug Abuse Screening Test-10 [Mean (Standard Deviation); unit: units on a scale] — DAST-10 total scores range from 0 to 10, with higher scores indicating more drug use related problems.
  units on a scale | 2.25 (2.06) | 1.58 (1.15) | 1.47 (1.52) | 1.71 (1.24) | 1.74 (1.52)
HIV status [Count of Participants; unit: Participants]
  HIV negative | 29 | 37 | 32 | 31 | 129
  HIV positive | 3 | 3 | 2 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Respondents Reporting Any Drug Use
Description: The outcome measure is a dichotomous variable indicating whether or not each participant reported any drug use in the in the 30 days prior to each follow-up assessment. The table below displays the number (and percentage) of participants who indicated the use of any drugs at each assessment wave. Assessments were conducted at 1, 3, and 6 month post intervention.
Time Frame: 30 days prior to assessment
Population: Intent to treat analysis conducted using latent growth curve modeling to examine between-group differences in follow-up rates of drug use and trajectories of use over the follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
Number analyzed (Participants) | 32 | 40 | 34 | 34
Participants
  1 month follow-up: number analyzed (Participants) | 29 | 37 | 32 | 31
  1 month follow-up | 25 | 26 | 18 | 17
  3 month follow-up: number analyzed (Participants) | 26 | 36 | 30 | 31
  3 month follow-up | 20 | 17 | 28 | 15
  6 month follow-up: number analyzed (Participants) | 25 | 37 | 28 | 31
  6 month follow-up | 15 | 31 | 15 | 17
Statistical Analysis 1: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = .03, multi-leve latent growth curve — A multi-level latent growth curve (LGC) with a intercept and linear slope was specified. The main effects of SUM and CT video were modeled at level 2 in addition to their interaction. Drug use was specified as a binomial distribution; Beta = -3.62, 95% CI 2-sided [-6.78 to -0.46] — For 1-Month Follow-Up, substance use module (SUM) among those who did not view CT Video
Statistical Analysis 2: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = .18, multi-level latent growth curve — A multi-level latent growth curve (LGC) with an intercept and linear slope was specified. The main effects of SUM and CT video were modeled at level 2 in addition to their interaction. Drug use was specified as a binomial distribution; Beta = -1.67, 95% CI 2-sided [-4.10 to 0.76] — 1-month follow-up, effect of SUM among those who did view the CT video
Statistical Analysis 3: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.75, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.35, 95% CI 2-sided [-2.50 to 1.80] — 1-month follow up, effect of CT video among those who completed the SUM
Statistical Analysis 4: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.14, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -2.30, 95% CI 2-sided [-5.37 to 0.77] — 1-Month follow up, effect of CT video among those who did not complete SUM
Statistical Analysis 5: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.013, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -2.79, 95% CI 2-sided [-5.00 to -0.58] — 3-Month follow up, effect of SUM among those who viewed the CT video
Statistical Analysis 6: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.10, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -2.09, 95% CI 2-sided [-4.56 to 0.38] — 3-Month follow up, effect of SUM among those who did not view CT video
Statistical Analysis 7: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; A multi-level latent growth curve (LGC) with an intercept and linear slope was specified. The main effects of SUM and CT video were modeled at level 2 in addition to their interaction. Drug use was specified as a binomial distribution; Test type: Superiority; p = 0.78, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = 0.40, 95% CI 2-sided [-2.35 to 3.16] — 3-month follow-up, effect of CT Video among those who completed the SUM
Statistical Analysis 8: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.75, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.30, 95% CI 2-sided [-2.12 to 1.53] — 3-month follow-up, effect of CT video among those who did not complete SUM
Statistical Analysis 9: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.014, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -3.93, 95% CI 2-sided [-7.06 to -0.81] — 6-month follow-up, effects of SUM among those who viewed the CT video
Statistical Analysis 10: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.67, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.57, 95% CI 2-sided [-3.16 to 2.03] — 6-month follow up, effect of SUM among those who did not view CT video
Statistical Analysis 11: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.83, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.24, 95% CI 2-sided [-2.39 to 1.91] — 6-month follow up, effect of CT video among those who completed the SUM
Statistical Analysis 12: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.05, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = 3.13, 95% CI 2-sided [-0.004 to 6.25] — 6-month follow-up, effects of CT video among those who did not complete SUM

2. Primary Outcome: Condomless Anal Sex With Casual Partners
Description: The outcome measure is a dichotomous variable indicating whether or not each participant indicated the occurrence of any insertive or receptive condomless anal sex (CAS) with a casual partner in the 30 days prior to each follow-up assessment. The table below displays the number (and percentage) of participants who indicated any CAS with a casual partner at each assessment wave. Assessments were conducted at 1, 3, and 6 month post intervention.
Time Frame: 30 days prior to assessment
Population: n reported is number retained at each wave
Measure: Count of Participants; unit: Participants
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
Number analyzed (Participants) | 32 | 40 | 34 | 34
Participants
  1 month follow-up: number analyzed (Participants) | 29 | 37 | 32 | 31
  1 month follow-up | 3 | 3 | 3 | 1
  3 month follow-up: number analyzed (Participants) | 26 | 36 | 30 | 31
  3 month follow-up | 0 | 5 | 6 | 2
  6 month follow-up: number analyzed (Participants) | 25 | 37 | 28 | 31
  6 month follow-up | 3 | 4 | 10 | 3
Statistical Analysis 1: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.90, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = 0.05, 95% CI 2-sided [-2.30 to 2.41] — Effect of SUM on the latent intercept factor among those who did not view CT videos
Statistical Analysis 2: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.78, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = 0.26, 95% CI 2-sided [-2.23 to 2.75] — Effects of CT video on the latent intercept factor among those who did not view SUM
Statistical Analysis 3: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.53, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -1.18, 95% CI 2-sided [-4.86 to 2.51] — Effects of the interaction between SUM and CT video on the latent intercept
Statistical Analysis 4: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.14, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = 1.83, 95% CI 2-sided [-0.62 to 4.29] — Effect of SUM on the latent slope factor among those who did not view CT Videos
Statistical Analysis 5: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.76, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = 0.35, 95% CI 2-sided [-2.02 to 2.72] — Effects of CT Video on latent slope factor among those who did not complete the SUM
Statistical Analysis 6: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.45, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -1.28, 95% CI 2-sided [-4.62 to 2.06] — Effects of the interaction between SUM and CT videos in the prediction of the latent slope factor

3. Primary Outcome: Drug Abuse Screening Test-10 Total Scores
Description: The scale assesses the number of drug use related problems experienced by the participant in the 30 days prior to the assessment. Higher scores indicate a greater number of drug use related problems. Note, assessments were conducted at 1, 3, and 6 months post intervention.
Time Frame: 30 days prior to assessment
Population: n reported is the number retained at each follow-up wave.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
Number analyzed (Participants) | 32 | 40 | 34 | 34
score on a scale
  1 month follow-up: number analyzed (Participants) | 29 | 37 | 32 | 31
  1 month follow-up | 2.52 (2.04) | 1.70 (1.75) | 1.16 (1.39) | 1.06 (1.18)
  3 month follow-up: number analyzed (Participants) | 26 | 36 | 30 | 31
  3 month follow-up | 1.98 (2.01) | 1.53 (1.42) | 1.40 (1.85) | 0.71 (0.90)
  6 month follow-up | 1.76 (2.12) | 1.70 (1.56) | 1.25 (1.73) | 0.84 (1.00)
Statistical Analysis 1: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.02, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.75, 95% CI 2-sided [-1.39 to -0.11] — 1-month follow-up, effect of SUM among those who viewed CT videos
Statistical Analysis 2: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.10, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.49, 95% CI 2-sided [-1.07 to 0.09] — 1-month follow-up, effect of SUM among those who did not view CT videos
Statistical Analysis 3: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.63, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.15, 95% CI 2-sided [-0.77 to 0.47] — 1-month follow-up, effects of CT video among those who completed SUM
Statistical Analysis 4: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.19, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.41, 95% CI 2-sided [-1.01 to 0.20] — 1-month follow-up, effects of CT video among those who did not complete SUM
Statistical Analysis 5: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.01, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.64, 95% CI 2-sided [-1.13 to -0.15] — 3-month follow-up, effect of SUM among those who completed the CT video
Statistical Analysis 6: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.12, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.49, 95% CI 2-sided [-1.11 to 0.12] — 3-month follow-up, effects of SUM among those who did not complete CT video
Statistical Analysis 7: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.23, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.34, 95% CI 2-sided [-0.89 to 0.21] — 3-month follow-up, effects of CT video among those who completed SUM
Statistical Analysis 8: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.51, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.19, 95% CI 2-sided [-0.76 to 0.38] — 3-month follow-up, effect of CT video among those who did not complete SUM
Statistical Analysis 9: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.003, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.79, 95% CI 2-sided [-1.32 to -0.27] — 6-month follow-up, effects of SUM among those who viewed CT videos
Statistical Analysis 10: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.49, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.25, 95% CI 2-sided [-0.96 to 0.46] — 6-month follow-up, effect of SUM among those who did not view the CT video
Statistical Analysis 11: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.10, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.53, 95% CI 2-sided [-1.16 to 0.11] — 6-month follow-up, effect of CT video among those who completed SUM
Statistical Analysis 12: Comparison: CHTC as Usual vs CHTC + Communication Skills Videos vs CHTC + Substance Use Module vs CHTC + Video + Substance Use Module; Test type: Superiority; p = 0.96, multi-level latent growth curve — [p-value comment as in outcome 1, analysis 2]; Beta = -0.02, 95% CI 2-sided [-0.60 to 0.64] — 6-month follow-up, effect of CT video among those who did not complete SUM

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for a period of 6 months from baseline to final assessment.
Arm/Group | CHTC as Usual | CHTC + Communication Skills Videos | CHTC + Substance Use Module | CHTC + Video + Substance Use Module
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/40 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/40 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/32 | 0/40 | 0/34 | 0/34

LIMITATIONS AND CAVEATS:
The design does not permit inferences about effects of components delivered independently of CHTC.

The sample was recruited in a major metropolitan area and at relatively lower risk for HIV infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03125915/Prot_SAP_000.pdf